CLINICAL TRIAL: NCT05285956
Title: Feasibility of Calm to Reduce Stress and Improve Sleep During Pregnancy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Personnel Change
Sponsor: Calm.com, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Calm2021-102
Record Dates: First submitted 2022-02-23; First posted 2022-03-18 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Pregnancy Related

STUDY DESIGN:
Masking Description: Researchers will assign participants to groups based on a randomized allocation list, which will be generated prior to the start study by a team member who is not involved in the group-assignment process. Allocation sequences will be concealed until the time of group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants (n=90) will be provided free access to and asked to register for the consumer-based mobile meditation app, Calm, on their phone. Participants will then receive an email containing one year of free access to Calm. Participants will be asked to use Calm at least 10 minutes per day for 8 weeks. Women will be asked to use 10 sessions of specific pregnancy content for the first four weeks and then will have autonomy to use the app how they prefer for the remainder of the study period (with continued encouragement to use the pregnancy meditations)
  Interventions: Behavioral: Calm app
- Control (No Intervention): Participants (n=90) will be asked to continue with usual care and complete survey measures at each time point.

INTERVENTIONS:
Behavioral: Calm app — Calm is a popular, subscription-based, meditation app accessible across web-based and smartphone platforms (iOS and Android) with over 100 million downloads and four million subscribers. The app offers a range of content rooted in mindfulness principles to help users incorporate mindfulness into their lives and generally promote wellbeing (e.g., a large library of guided meditations including the 10-minute Daily Calm, Sleep Stories, educational courses, mindful movement, music, and nature scenes and sounds). Calm also teaches users the basics of mindfulness, includes components to remind users to meditate, track user activity, and allow users to share their status with others. The feasibility of the app and its efficacy for improving mental health outcomes (i.e., stress, anxiety, and depressive symptoms), mindfulness, and sleep have been previously tested in various populations providing evidence that using Calm may improve wellbeing.
  Arms: Intervention

SUMMARY:
Purpose: Test the effects of using Calm for its impact on stress, anxiety, and sleep in pregnant women using the following aims:

Aim #1: Determine the feasibility of using Calm.

Aim #2: Determine the preliminary efficacy of using Calm on stress, anxiety, and sleep.

Exploratory Aim #3: Explore the preliminary efficacy of using Calm on self-reported birth outcomes

DETAILED DESCRIPTION:
Rates of stress and poor sleep affect up to 70% of pregnant women with rates even higher in racial and ethnic minority (REM) women. Stress and poor sleep are often untreated or misdiagnosed, especially in lower income and REM populations, due to high health-related costs or lack of insurance and may underestimate the prevalence of stress and poor sleep. High stress and poor sleep increases risk of depression, anxiety, pregnancy complications, and poor birth outcomes. Research suggests that stress and poor sleep are strongly associated during pregnancy. In fact, poor sleep in pregnancy has been regarded as both an outcome of stress and a stressor in itself and improving sleep has been suggested as a strategy to protect maternal mental health. There is a need for interventions particularly among REM pregnant women to reduce stress and improve sleep.

Treatments for prenatal stress and poor sleep are inadequate in meeting the needs of pregnant women. Typical treatments are usually an aggregation of medication, interpersonal psychotherapy, and cognitive behavioral therapy. However, mental health stigma and concern with potential teratogenic effects from medication use may discourage women to seek help and many prefer non-pharmacological approaches. Mindfulness meditation (MM) is a nonpharmacological approach effective for reducing stress and improving sleep during pregnancy. MM can be described as the practice of self-regulation of attention and accepting the present moment. MM interventions may moderate the impact of poor sleep quality on stress and can have lasting effects with regular practice. Furthermore, MM is a recommended strategy for pregnant women to improve mental health. While there is evidence for the benefits of MM, many studies report high drop-out rates due to inconvenience, travel, or child care demands. Accessible, low cost, MM interventions to improve stress and sleep outcomes for pregnant women are warranted.

Delivery of MM using smartphone applications (apps) for the management of stress and sleep has dramatically increased in recent years. App-based MM can be delivered remotely, substantially increasing reach, accessibility, and scalability. Over 260 MM apps exist, but many consumer-based apps have low evidence for their efficacy among pregnant and REM users. Calm is a popular, consumer-based MM app that has over 100 million downloads, four million subscribers, and has demonstrated effects in stress and improved sleep in non-pregnant populations. In our preliminary survey data, pregnant subscribers of the Calm app most commonly used the app for sleep problems (29%; n=31) and reported the app was most helpful for improving sleep (32%; n=32) and stress (21%; n=21). Currently, the feasibility and potential impact of the Calm app to reduce stress and improve sleep in pregnant REM women is unknown.

ELIGIBILITY:
Inclusion Criteria

* Pregnant women 14-16 or 28-30 weeks gestation
* Resident of United States
* Access to regular WiFI
* Access to a smartphone regularly
* Willing to download an app onto their smartphone
* Score of >13 on Perceived Stress Scale (PSS-10)] 31 and sleep quality [score of >5 on Pittsburgh Sleep Quality Index (PSQI)]
* Have not practiced meditation more than 60 minutes a month in the past six months
* Willing to be randomized to one of two groups.

Exclusion Criteria:

* <18 years of age
* Unable to consent
* First trimester (less than 14 weeks)

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 4 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Change in Stress (Perceived Stress Scale) | Baseline, 4 weeks, 8 weeks
  The Perceived Stress Scale (PSS) is a 10-item scale. Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress. Scores ranging from 0-13 would be considered low stress. Scores ranging from 14-26 would be considered moderate stress. Scores ranging from 27-40 would be considered high perceived stress.
Change in Sleep Quality (Pittsburgh Sleep Quality Index) | Baseline, 4 weeks, 8 weeks
  The Pittsburgh Sleep Quality Index (PSQI) contains 19 self-rated questions. The items are combined to form seven "component" scores, each of which has a range of 0-3 points. In all cases, a score of "0" indicates no difficulty, while a score of "3" indicates severe difficulty. The seven component scores are then added to form one "global" score, with a range of 0-21, "0" indicating no difficulty, and "21" indicating severe difficulties in all areas.
Change in Depressive Symptoms (Edinburgh Postnatal Depression Scale) | Baseline, 4 weeks, 8 weeks
  The 10-question Edinburgh Postnatal Depression Scale (EPDS) is a valuable, efficient, and proven effective screening tool for identifying patients at risk for "perinatal" depression. Mothers who score above 13 are likely to be suffering from a depressive illness of varying severity. The scale indicates how the mother has felt during the previous week.
Change in Anxiety (Pregnancy Related Anxiety Questionnaire) | Baseline, 4 weeks, 8 weeks
  The Pregnancy Related Anxiety Questionnaire, Revised version 2 (PRAQ-R2 ) contains 10 questions, grouped into three subscales: fear of giving birth (FoGB; items 1, 2, and 6), worries of bearing a physically or mentally handicapped child (WaHC; items 4, 9, 10, and 11); and concern about own appearance (CoA; items 3, 5, and 7). An additional item is ("I am anxious about the delivery"). The total score (ranging from 10 to 50 points) and the sum of item scores that make up the three subscales are calculated. Higher scores are assumed to indicate increased pregnancy related anxiety intensity. No clinical cutoff point is currently defined for this tool.

SECONDARY OUTCOMES:
Self-Reported Baby's Gestational Age at Birth | 2 weeks post due date
  Gestational age
Self-Reported Baby's Birth Weight | 2 weeks post due date
Self-reported Childbirth Experience | 2 weeks post due date
  Childbirth Experience Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jen Huberty, PhD, Study Director — Calm.com, Inc.
Locations (1):
- Calm, Inc., San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huberty J, Puzia ME, Green J, Vlisides-Henry RD, Larkey L, Irwin MR, Vranceanu AM. A mindfulness meditation mobile app improves depression and anxiety in adults with sleep disturbance: Analysis from a randomized controlled trial. Gen Hosp Psychiatry. 2021 Nov-Dec;73:30-37. doi: 10.1016/j.genhosppsych.2021.09.004. Epub 2021 Sep 11. PMID 34537477
- [Background] Huberty JL, Green J, Puzia ME, Larkey L, Laird B, Vranceanu AM, Vlisides-Henry R, Irwin MR. Testing a mindfulness meditation mobile app for the treatment of sleep-related symptoms in adults with sleep disturbance: A randomized controlled trial. PLoS One. 2021 Jan 7;16(1):e0244717. doi: 10.1371/journal.pone.0244717. eCollection 2021. PMID 33411779
- [Background] Huberty J, Puzia ME, Larkey L, Irwin MR, Vranceanu AM. Use of the Consumer-Based Meditation App Calm for Sleep Disturbances: Cross-Sectional Survey Study. JMIR Form Res. 2020 Nov 13;4(11):e19508. doi: 10.2196/19508. PMID 33185552
- [Background] Huberty J, Green J, Glissmann C, Larkey L, Puzia M, Lee C. Efficacy of the Mindfulness Meditation Mobile App "Calm" to Reduce Stress Among College Students: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2019 Jun 25;7(6):e14273. doi: 10.2196/14273. PMID 31237569
- [Background] Kwok OM, Underhill AT, Berry JW, Luo W, Elliott TR, Yoon M. Analyzing Longitudinal Data with Multilevel Models: An Example with Individuals Living with Lower Extremity Intra-articular Fractures. Rehabil Psychol. 2008 Aug;53(3):370-386. doi: 10.1037/a0012765. PMID 19649151
- [Background] Gravel J, Opatrny L, Shapiro S. The intention-to-treat approach in randomized controlled trials: are authors saying what they do and doing what they say? Clin Trials. 2007;4(4):350-6. doi: 10.1177/1740774507081223. PMID 17848496